CLINICAL TRIAL: NCT01668706
Title: Pharmacogenomics Study of Sleep Disturbance and Neurocognitive Impairments in the Opioid Addicts
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: MD098SCW01
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2012-08

CONDITIONS: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, DNA and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Methadone maintenance treatment (MMT)
- Buprenorphine-Naloxone treatment (BNT)
- Medication-free ex-addicts(MF)
- Normal control (NC)

SUMMARY:
Opioid abuse is a complex problem, which not only impacts on addicts' physical and psychological health individually, but also threats the society. Recently, spread of HIV via sexual behavior and needle sharing among injecting drug users (IDUs) also becomes a serious public health problem all over the world. In Taiwan, since the first HIV-infected IDU identified in 1987, the incident cases have mounted to 2,461 in 2005. To prevent the epidemics of HIV among IDUs, the Center for Disease Control (CDC) thus collaborated with Department of Justice and implemented harm reduction programs in 2005. It is the milestone that opioid addiction is officially treated as a health rather than a legal issue in Taiwan. Among the harm reduction programs of needle and syringe exchange for IDUs as well as substitution treatment for opioid dependence, methadone maintenance treatment (MMT) is one of the most important parts. Till 2008, there were over 13,000 heroin addicts participated in more than 80 MMT programs.

Although the clinical evidences have proven the superior effectiveness of maintenance therapy in ameliorating illicit substances abuse, decreasing criminality and improving quality of life, there are common problems of sleep disturbance and neurocognitive impairments among the subjects receiving opioid medications. The concerns of the adverse effects might thus frustrate the subjects' motivation and compliance to maintain treatments. However, sleep disturbance and neurocognitive impairments related to opioid medications are often neglected in the clinical practices and there are scanty researches focusing on these crucial issues in the existing literature.

In this prospective study, four groups of subjects including methadone maintenance treatment, buprenorphine/naloxone, medication-free opioid ex-addicts and healthy volunteers will be enrolled. Via the comprehensive assessments including clinical interview, neurocognitive examinations, electrocardiogram-based sleep breathing detector and pharmacogenomical evaluation, we will not only have the opportunities to have more insights on the impacts of opioid medications on sleep and neurocognitive performances, but also develop more adequate strategies to improve motivation and outcome in treating the opioid addicts.

ELIGIBILITY:
1. Normal control group (NC):

   Inclusion criteria:
   1. Chinese ethnicity
   2. Men or women above age of 20
   3. Able to participate in a clinical assessment in Chinese (including Mandarin and Taiwanese dialects)
   4. Individuals who have completed a written consent form

   Exclusion criteria:
   1. Patients with comorbid severe mental disorders including:

      1. Organic mental disorders, or
      2. Schizophrenia
   2. Past diagnosis of Heroin dependence by DSM-IV definition
   3. Severe cognitive impairment
   4. Being pregnant
2. Methadone maintenance treatment group (MMT)

   Inclusion criteria:
   1. Chinese ethnicity
   2. Men or women above age of 20, below age of 65
   3. Able to participate in a clinical assessment in Chinese (including Mandarin and Taiwanese dialects)
   4. Diagnosis of Heroin dependence by DSM-IV definition
   5. Enter methadone maintenance therapy for at least 3 months
   6. No change of methadone dosage for the last week
   7. Regularly took methadone for the last week
   8. Individuals who have completed a written consent form

   Exclusion criteria:
   1. Patients with comorbid severe mental disorders including:

      1. Organic mental disorders, or
      2. Schizophrenia
   2. Severe cognitive impairment
   3. Being pregnant
3. Buprenorphine/Naloxone treatment group (BNT)

   Inclusion criteria:
   1. Chinese ethnicity
   2. Men or women above age of 20, below age of 65
   3. Able to participate in a clinical assessment in Chinese (including Mandarin and Taiwanese dialects)
   4. Diagnosis of Heroin dependence by DSM-IV definition
   5. Enter buprenorphine maintenance therapy for at least 3 months
   6. No change of buprenorphine dosage for the last week
   7. Regularly took buprenorphine for the last week
   8. Individuals who have completed a written consent form

   Exclusion criteria:
   1. Patients with comorbid severe mental disorders including:

      1. Organic mental disorders, or
      2. Schizophrenia
   2. Severe cognitive impairment
   3. Being pregnant
4. Medication-free ex-addict group (MF)

Inclusion criteria:

1. Chinese ethnicity
2. Men or women above age of 20
3. Able to participate in a clinical assessment in Chinese (including Mandarin and Taiwanese dialects)
4. Diagnosis of Heroin dependence by DSM-IV definition
5. Individuals who have completed a written consent form

Exclusion criteria:

1. Patients with comorbid severe mental disorders including:

   1. Organic mental disorders, or
   2. Schizophrenia
2. Severe cognitive impairment
3. Being pregnant
4. Exposure of methadone, buprenorphine and other opioid treatment in the previous 3 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal control group:
     Healthy adults will be recruited from community.
  2. Methadone Maintenance treatment group Study subjects will be enrolled only in the methadone clinic.
  3. Buprenorphine/Naloxone treatment group Subjects will be enrolled only in the clinic.
  4. Drug-free ex-addict group Subjects will be recruited from the therapeutic communities and halfway house of Operation Dawn.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Group differences in demopraphics | one year
  support system, vital sign, substance use history

SECONDARY OUTCOMES:
Gruop differences in neuro-cognitive functions | one year
  attention, executive function, decision making

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chang Wang, M.D., M.Sc., Principal Investigator — National Health Research Institutes, Taiwan
Locations (5):
- Taiwan (5):
  - ChangHua Christian Hospital, Lukang, ChangHua
  - Far Eastern Memorial Hospital, Banqiao District, New Taipei City
  - Far Eastern Memorial Hospital, Banqiao District, New Taipei
  - En-Chu-Gong Hospital, Sanxia District, New Taipei
  - National Health Research Institute, Miaoli County, Taiwan